CLINICAL TRIAL: NCT06798129
Title: Effects of Extracorporeal Treatment in Patients With Acute Poisoning in Jiangsu Province, China: A Multi-center Target Trial Emulation
Brief Title: Effects of Extracorporeal Treatment in Patients With Acute Poisoning
Status: Active, not recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, MD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2025-1054-01-01
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Poisoning; Extracorporeal Treatment
MeSH Terms: conditions — Poisoning | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Extracorporeal Treatment — Extracorporeal treatments include hemoperfusion, hemodialysis, continuous kidney replacement therapy, and plasma exchange.

SUMMARY:
This study aims to estimate the effect of extracorporeal treatments (ECTRs) on 28-day survival in patients with acute poisoning. The treatment strategy was receipt of ECTR (hemoperfusion, hemodialysis, continuous kidney replacement therapy, and/or or plasma exchange) versus a non-ECTR strategy.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age and older
* History of acute poisoning

Exclusion Criteria:

* missing records in survival outcome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with acute poisoning
Sampling Method: Non-Probability Sample
Enrollment: 5269 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival outcome | 28 days within the index date of presentation at emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China